CLINICAL TRIAL: NCT01360723
Title: Comparison of DNA Methylation Between Urothelial Carcinoma and Healthy Controls
Brief Title: DNA Methylation and Arsenic-associated Urothelial Carcinoma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: China Medical University Hospital (Other)
Responsible Party: Chi-Jung Chung and Chao-Hsian Chang, Department of Urology
Other Study IDs: DMR100-IRB-080
Record Dates: First submitted 2011-05-24; First posted 2011-05-26 (Estimated); Last update posted 2011-05-27 (Estimated); Status verified 2011-05

CONDITIONS: Urothelial Carcinoma
MeSH Terms: conditions — Carcinoma, Transitional Cell

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- urothelial carcinoma: Pathological verification of UC was done by routine urological practice including endoscopic biopsy or surgical resection of urinary tract tumors followed by histopathological examination by board-certified pathologists.
- Healthy controls group: Age and gender matched control subjects with no evidence of UC or any other malignancy were accrued from the hospital, recruiting people receiving adult health examinations at China Medical University Hospital.

SUMMARY:
The investigators previously pointed out the significant association between urinary arsenic profiles and urothelial carcinoma (UC) risk through a 12-year follow-up study. Further, the investigators observed the increased UC risk in people with lower plasma folate and higher homocysteine than those with higher plasma folate and lower homocysteine in 2010. S-adenosylmethionine (SAM) is one factor included in one-carbon metabolism pathway and is the main donor of methyl group in cells. The ratio of SAM and its metabolite S-adenosylhomocysteine (SAH) not only reflected the intake level of dietary folate but also demonstrated the extent of global DNA methylation. These factors might play important roles in UC carcinogenesis. The investigators would expect to take three years to explore the interactions among global DNA methylation, one-carbon metabolic pathway factors, urinary arsenic profiles, the polymorphisms and haplotype of Glycine N-methyltransferase (GNMT) and UC. In the first year, the investigators would measure the levels of plasma folate, homocysteine, SAM and SAH and evaluate the associations between these factors and UC risk. In the second year, the investigators would set up the method of immunohistochemistry stain and compare the differences between the global DNA methylation from bladder tissues and blood. In the last year, this investigators would analyze the GNMT gene polymorphism and haplotype variation. At the same time, the investigators would explore the impact of GNMT genetic variation and global DNA methylation on UC risk. Based on the results from our research, the investigators might propose that the decreased ratio of SAM/SAH resulted in UC risk increased. This mechanism might be through the changed levels of urinary arsenic profiles and global DNA methylation.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of urothelial carcinoma
* The voluntary of participating the study

Exclusion Criteria:

* Age smaller than 20 years
* Pregnant women
* Not willing to participate the study because of their personal reasons

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This is a hosital-based case-control study. Patients with urothelial carcinoma are recruited by pathological verification of UC was done by routine urological practice including endoscopic biopsy or surgical resection of urinary tract tumors followed by histopathological examination by board-certified pathologists. Healthy controls without evidence of UC or any other malignancy were recurited including those receiving adult health examinations at China Medical University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2011-05; Primary Completion 2014-05 (Estimated)

PRIMARY OUTCOMES:
urothelial carcinoma | up to three years

CONTACTS AND LOCATIONS:
Overall Officials: Chi-Jung Chung, PhD, Principal Investigator — Department of Health risk Management, China Medical University
Locations (1):
- Department of Urology, China Medical University Hospital, Taichung, Taiwan